CLINICAL TRIAL: NCT00465725
Title: A Randomized Crossover Oral Bioavailability Study Comparing the Pharmacokinetics and Pharmacodynamics of Picoplatin Administered Orally With Picoplatin Administered Intravenously in Subjects With Advanced Non-Hematological Malignancies
Brief Title: A Study Comparing Oral Picoplatin With Intravenous Picoplatin in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Poniard Pharmaceuticals (Industry)
Responsible Party: Robert Earhart, MD, PhD Study Director, Poniard Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0602 Oral Picoplatin
Record Dates: First submitted 2007-04-23; First posted 2007-04-25 (Estimated); Last update posted 2009-09-24 (Estimated); Status verified 2009-09

CONDITIONS: Bladder Cancer; Breast Cancer; Colorectal Cancer; Gastrointestinal Neoplasm; Head and Neck Cancer; Lung Cancer; Ovarian Cancer; Pancreatic Cancer; Prostate Cancer
Keywords: Picoplatin; tumor; cancer; sarcoma; neoplasm; advanced; platinum; chemotherapy; Solid Tumor
MeSH Terms: conditions — Urinary Bladder Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Gastrointestinal Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms; Neoplasms; Sarcoma | interventions — amminedichloro(2-methylpyridine)platinum(II)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): two-period crossover, open label study in which a single dose (Cycle 1) of picoplatin will be given either IV or PO, followed 4 weeks later by a single dose (Cycle 2) of picoplatin given by the route not used for Cycle 1. Subjects subsequently may continue to receive IV picoplatin commencing with Cycle 3 in a Continuation Study.
  Interventions: Drug: Picoplatin

INTERVENTIONS:
Drug: Picoplatin — The IV dose will be 120 mg/m2. Three oral dose levels will be studied sequentially (6 subjects per dose level) in the absence of dose limiting toxicity 200 mg, 300 mg, or 400 mg total dose.

SUMMARY:
Picoplatin is a new platinum-based chemotherapy drug that has been studied in a variety of cancers. Phase 1 and 2 studies have demonstrated that picoplatin may be effective in patients whose cancer returns or does not improve after treatment with chemotherapy. In these studies, picoplatin was administered intravenously. A capsule containing picoplatin has been formulated. This study will investigate the activity of the oral capsule in humans. Participants with advanced solid tumors will be enrolled.

DETAILED DESCRIPTION:
The primary study design is a randomized, two-period crossover, open label study in which a single dose (Cycle 1) of picoplatin will be given either IV or by oral capsule, followed 4 weeks later by a single dose (Cycle 2) of picoplatin given either IV or by oral capsule (whichever route was not used in Cycle 1). Participants may continue to receive cycles of IV picoplatin every 3 weeks, beginning with Cycle 3, as part of a Continuation Study.

This study will determine the relative safety, bioavailability, pharmacokinetics, pharmacodynamics, and urinary excretion of picoplatin administered orally with reference to picoplatin administered intravenously.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of non-hematological malignancy.
* Patients for whom no standard therapy exists and for whom, in the opinion of the investigator, treatments with single agent picoplatin is appropriate.
* 18 years of age or older.
* ECOG performance status 0-2.
* Life expectancy of at least 12 weeks.

(Additional inclusion criteria apply.)

Exclusion Criteria:

* Symptomatic or uncontrolled brain metastases.
* Prior radiation involving ≥ 30% of the total bone marrow space.
* Any concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study.
* Gastrointestinal surgery that might interfere with absorption of orally administered drug.
* Active inflammatory bowel disease, gastritis, ulcers, gastrointestinal or rectal bleeding.
* Clinical evidence of pancreatic injury or active pancreatitis.
* Female subjects who are pregnant or breastfeeding.

(Additional exclusion criteria apply.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2007-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
MTD | MTD
Comparison of platinum levels excreted in urine from 0-8 and 8-24 hours after start of IV or oral drug | PK

CONTACTS AND LOCATIONS:
Overall Officials: Robert Earhart, MD, PhD, Study Director — Poniard Pharmaceuticals
Locations (3):
- United States (3):
  - Georgia Cancer Specialists, Atlanta, Georgia
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Northwest Medical Specialties, Tacoma, Washington

REFERENCES:
- [Background] Beale P, Judson I, O'Donnell A, Trigo J, Rees C, Raynaud F, Turner A, Simmons L, Etterley L. A Phase I clinical and pharmacological study of cis-diamminedichloro(2-methylpyridine) platinum II (AMD473). Br J Cancer. 2003 Apr 7;88(7):1128-34. doi: 10.1038/sj.bjc.6600854. PMID 12671715
- [Background] Holford J, Raynaud F, Murrer BA, Grimaldi K, Hartley JA, Abrams M, Kelland LR. Chemical, biochemical and pharmacological activity of the novel sterically hindered platinum co-ordination complex, cis-[amminedichloro(2-methylpyridine)] platinum(II) (AMD473). Anticancer Drug Des. 1998 Jan;13(1):1-18. PMID 9474239
- [Background] Raynaud FI, Boxall FE, Goddard PM, Valenti M, Jones M, Murrer BA, Abrams M, Kelland LR. cis-Amminedichloro(2-methylpyridine) platinum(II) (AMD473), a novel sterically hindered platinum complex: in vivo activity, toxicology, and pharmacokinetics in mice. Clin Cancer Res. 1997 Nov;3(11):2063-74. PMID 9815598
- See also: Poniard Pharmaceuticals, Inc. — http://www.poniard.com